CLINICAL TRIAL: NCT03170583
Title: SJM Brady MRI Post Approval Study
Acronym: Brady MRI PAS
Status: Terminated | Type: Observational
Why Stopped: Abbott received FDA approval to transition the ongoing Brady MRI PAS study to EP a new EP-Passion Real World Evidence methodology
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP- CL1000304
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Bradycardia
Keywords: bradycardia, pacemaker, MRI scan
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: St. Jude Medical Tendril MRI™ lead — pacemaker, leads
  Other Names: St. Jude Medical Accent MRI™ pacemaker; St. Jude Medical Assurity MRI™ pacemaker; St. Jude Medical Endurity MRI™pacemaker

SUMMARY:
The purpose of this post approval study is to evaluate the long-term safety of the FDA approved St. Jude Medical Tendril MRI™ lead implanted with a SJM Brady MRI implantable pulse generator (IPG) such as the Accent MRI™, Assurity MRI™, Endurity MRI™ pacemaker, or similar model (SJM Brady MRI System) in subjects with a standard bradycardia pacing indication.

DETAILED DESCRIPTION:
This is a prospective, multi-center clinical study designed to evaluate the long-term safety of the Tendril MRI™ lead implanted with any SJM Brady MRI pacemaker or similar model (SJM Brady MRI system) in subjects with a standard bradycardia pacing indication through 60 months of follow up.

Additionally, the study will assess the safety of the pacemaker system in subject(s) undergoing clinically indicated MRI scan(s). Any enrolled subject implanted with the SJM Brady MRI system may be included in this evaluation if they are scheduled for or planning to have a MRI scan during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide informed consent for study participation (legally authorized representative is NOT acceptable).
2. Subject is at least 18 years of age or of legal age to give informed consent specific to state and national law.
3. Subject meets at least one of the following criteria:

   1. Is an Accent MRI IDE study subject who is being rolled over into the SJM Brady MRI PAS and still has at least one Tendril MRI™ lead implanted with a SJM Brady MRI pacemaker such as the Accent MRI or similar model.
   2. Is a subject who has been implanted with at least one Tendril MRI lead and a SJM Brady MRI pacemaker such as the Accent MRI or similar model, but is not part of the Accent MRI IDE study and will be enrolled within 30 days after implant.
   3. Is a subject who will be implanted with at least one Tendril MRI lead and a SJM Brady MRI pacemaker such as the Accent MRI or similar model and will be consented either at or within 30 days before implant.
4. Subject is willing and able to comply with the prescribed follow-up tests and schedule of evaluations including MRI scan procedures.

Exclusion Criteria:

1. Subject has been enrolled or intends to participate in a clinical drug and/or device study with an active treatment arm or that has any procedures, which could confound the results of this trial.
2. Subject is not expected to be able to complete the study follow up schedule or duration due to any health condition such as has malignancy, is deemed a candidate for transplant or Ventricular Assist Device, or in hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a standard bradycardia indication.
Sampling Method: Probability Sample
Enrollment: 1768 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from Tendril MRI RA lead-related complications through 60 months of follow up | 60 months
Freedom from Tendril MRI RV lead-related complications through 60 months of follow up | 60 months
MRI scan related complications rate through one-month following the MRI scan | 1 month

SECONDARY OUTCOMES:
The complication rate of the Tendril MRI lead | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, MS, Study Director — Abbott (formerly St. Jude Medical)
Locations (66):
- United States (66):
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Cardiology Associates of North East Arkansas, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mercy Hospital Northwest Arkansas, Rogers, Arkansas
  - Central Cardiology, Bakersfield, California
  - Raymond Schaerf, MD, Burbank, California
  - St. Helena Hospital, Deer Park, California
  - USC University Hospital, Los Angeles, California
  - Riverside Medical Clinic, Riverside, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - San Diego Heart Rhythm Center, San Diego, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Shands Jacksonville, Jacksonville, Florida
  - Hrachian Hakop MD PA, South Miami, Florida
  - Cardiology Partners, Wellington, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Atlanta Heart Specialist, Cumming, Georgia
  - Coliseum Medical Centers, Macon, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - MidMichigan Medical Center-Midland, Midland, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Missouri Heart Center, Columbia, Missouri
  - St. Luke's Hospital, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Kearney Regional Medical Center, Kearney, Nebraska
  - BryanLGH Medical Center East, Lincoln, Nebraska
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New Brunswick Cardiology Group, Somerset, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Capital Cardiology Associates, Albany, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Hudson Valley Cardiovascular Practice, P.C., Poughkeepsie, New York
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Abington Medical Specialists, Abington, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - BCS Heart, LLP, College Station, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Fort Worth Heart, Fort Worth, Texas
  - Houston Cardiovascular Associates, Houston, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Carient Heart & Vascular, P.C., Manassas, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Medical Group, Milwaukee, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
  - Cheyenne Cardiology Associates, Cheyenne, Wyoming